CLINICAL TRIAL: NCT07118033
Title: Evaluation of the Specificity of a Manual Therapy Based on a Decision Algorithm (Algo-K) in the Physiotherapy Treatment of Sub Acute Low Back Pain With Radiating Pain
Brief Title: Algo K Specific Manual Therapy for Sub Acute Low Back Pain With Radicular Symptoms
Acronym: ALGO-K
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: APHP230858; 2024-A01892-45 (Other: IDRCB)
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Sub Acute Low Back Pain With Radiating Symptoms
Keywords: Low back pain; Manual therapy; Physiotherapy; Decision making
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: 2 groups, both of them will execute the same standard physiotherapy care based on exercise and education for 25 minutes for each session, randomly assigned 1:1.
  For the control group, they will have a 5 minutes postero-anterior mobilisation procedure on a upper thoracic vertebra For the interventional group, they will have a 5 minutes postero-anterior mobilisation procedure on a lumbar vertebra, determined by the algorithm
Who Masked: Participant
Masking Description: Patients unaware of allocation ; sham mobilization in control arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Specific manual therapy (Experimental): Usual exercise based physiotherapy + 5 min lumbar PA mobilisations chosen with Algo K algorithm based on symptom response
  Interventions: Procedure: Specific Manual Therapy
- Non specific manual therapy (Sham Comparator): Same physiotherapy + 5 min PA mobilisations in upper thoracic spine, distant from symptoms
  Interventions: Procedure: Non specific Manual Therapy

INTERVENTIONS:
Procedure: Specific Manual Therapy — Participants in this group receive a standardized physiotherapy program (exercise and education) plus 5 minutes of targeted lumbar postero anterior mobilizations. These mobilizations are selected using the Algo K decision algorithm, which guides the therapist to choose the most appropriate technique based on the patient's pain response during preliminary movement tests.
  Arms: Specific manual therapy
Procedure: Non specific Manual Therapy — Participants in this group receive the same physiotherapy program, but the additional 5 minutes of mobilization are applied to the upper thoracic spine (T4-T7), away from the symptomatic lumbar region. This sham mobilization mimics the manual therapy without targeting the affected area or following the algorithm's logic.
  Arms: Non specific manual therapy

SUMMARY:
This study evaluates the effectiveness of a specific manual therapy approach based on the Algo-K decision algorithm in patients with subacute low back pain radiating to the lower limb. Algo-K helps select the most suitable lumbar mobilization technique according to the patient's pain response. The experimental group will receive a five-minute targeted manual therapy in addition to standard physiotherapy, while the control group will receive a non-specific mobilization. The study aims to determine whether this algorithm-guided intervention leads to faster and greater improvement in pain and disability.

DETAILED DESCRIPTION:
Subacute low back pain (LBP) with radiating symptoms is a common musculoskeletal disorder with a risk of chronicization. Manual therapy is often used in physiotherapy to treat LBP, but its effectiveness varies widely due to heterogeneous practices and lack of specificity. The Algo-K algorithm was developed to guide therapists in selecting the most appropriate mobilization technique based on patients' symptomatic responses during movement tests.

This multicenter randomized controlled trial compares the effectiveness of a specific manual therapy guided by the Algo-K algorithm versus a non-specific manual therapy added to a standardized exercise-based physiotherapy program. Sixty adult patients with subacute LBP and radiating pain will be included. Participants will be randomly assigned to either:

* Experimental group: 5 minutes of specific lumbar mobilizations based on the Algo-K decision tree;
* Control group: 5 minutes of non-specific mobilization at a distant thoracic level.

Both groups will receive the same standard physiotherapy care based on exercise and education, delivered over 12 sessions within a 60-day period.

The primary outcome is the Oswestry Disability Index (ODI) score at 26-30 days. Secondary outcomes include pain intensity (Numeric Rating Scale), pain distribution (body diagram), and long-term disability (ODI at 52-60 days). The hypothesis is that the specific, patient-tailored manual therapy will improve functional outcomes and reduce pain more effectively than non-specific mobilization.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 65 y o
* Sub acute low back pain (7 days - 3 months) with irradiation to one lower limb, pain 3 10/10
* Mechanically responsive pain
* ODI > 20 % and < 80 %
* Prescription ≥ 12 physiotherapy sessions (or un specified)
* Able to complete 12 sessions in ≤ 60 days
* Affiliated to French social security
* Signed informed consent

Exclusion Criteria:

* Suspicion or history of serious pathology (cancer, systemic inflammatory disease, etc.)
* Main complaint other than low back pain with irradiation
* Prior spine or hip surgery (no time limit) / thoraco abdominal surgery < 3 y
* Central Sensitization Inventory ≥ 37
* HAD anxiety or depression sub score ≥ 8
* Planned lumbar infiltration during follow up
* Pregnancy or breastfeeding
* Legal protection (guardianship, custody, imprisonment)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI, %) | Baseline day to 26-30
  Patient-reported disability (ODI French version)

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI, %) | day 52-60 /or visit 12
  Disability at end of follow-up
Pain intensity (numeric rating scale, 0-10) | Baseline day 26-30 ; day 52-60 /or visit 12
  Average pain last 24h
Pain topography (body diagram score) | Baseline day 26-30 ; day 52-60 /or visit 12
  Distal extension of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: valerie VACHER, Study Chair — DRCI-AP-HP, Saint-Louis Hospital

IPD SHARING:
Plan to Share IPD: No